CLINICAL TRIAL: NCT06300411
Title: A Phase 1 Study of SRG-514 Administered Intraoperatively to the Site of Tumor Resection of Patients Undergoing Breast-Conserving Cancer Surgery
Brief Title: SRG-514 Administered Intraoperatively to Patients Undergoing Breast-conserving Cancer Surgery
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: SURGE Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SRG-514-01
Record Dates: First submitted 2024-03-01; First posted 2024-03-08 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: Intraoperative; Ketorolac; Open-label; SRG-514; Dose escalation; Immunotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SRG-514 (Experimental): SRG-514
  Interventions: Drug: SRG-514

INTERVENTIONS:
Drug: SRG-514 — SRG-514 monotherapy

SUMMARY:
This is a multicenter, first-in-human (FIH), open label, Phase 1 dose escalation and recommended Phase 2 dose (RP2D) extension trial with a primary objective to define the RP2D of SRG-514 when administered intraoperatively to patients undergoing breast-conserving cancer surgery. SRG-514 will be investigated utilizing a 3+3 convention dose escalation cohorts.

DETAILED DESCRIPTION:
This is a multicenter, first-in-human (FIH), open label, Phase 1 dose escalation and recommended Phase 2 dose (RP2D) extension trial with a primary objective to define the RP2D of SRG-514 when administered intraoperatively to patients undergoing breast-conserving cancer surgery. SRG-514 will be investigated utilizing a 3+3 convention dose escalation cohorts, with 3 to 6 patients enrolled at each dose level, and a minimum of 6 patients enrolled at the highest dose level, for a total of approximately 12-18 patients in the dose escalation portion of the study.

SRG-514 doses will be escalated based on safety and potential dose-limiting toxicities (DLTs) within the 14-day period following SRG-514 administration. Patients who do not complete the DLT period for reasons other than study drug related toxicity would be considered non-evaluable for DLT assessment and may be replaced.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Body weight >50kg
* Have a history of histologically confirmed diagnosis of breast carcinoma or ductal carcinoma in situ, except inflammatory breast cancer.
* Plan to undergo breast-conserving surgical treatment of breast cancer with curative intent. Adjuvant or neoadjuvant chemotherapy is allowed.
* Have Eastern Cooperative Oncology Group (ECOG) Performance Status <2
* Have adequate organ and bone marrow function at screening

Exclusion Criteria:

* Any known contraindication to ketorolac or other non-steroidal anti-inflammatory drugs (NSAIDs)
* Patients anticipated to require the use of a drain after breast-conserving surgery (BCS)
* Patients undergoing immediate reconstruction surgery, intraoperative radiation therapy (IORT) or brachytherapy requiring the placement of balloons or catheters during the lumpectomy procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) [Safety and Tolerability] | 14 days
  Incidence of dose-limiting toxicities (DLTs) over the first 14-days of study treatment
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Time on trial up to 60 days
  Incidence of serious adverse events (SAEs), and adverse events (AEs), graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0

SECONDARY OUTCOMES:
Pharmacokinetics of SRG-514 | Day 0, Day 1, Day 2
  Maximum plasma concentration (Cmax) of ketorolac in patient blood
Pharmacokinetics of SRG-514 | Day 0, Day 1, Day 2
  Area under the plasma concentration versus time curve (AUC) of ketorolac in patient blood
Pharmacodynamics of SRG-514 | Day 0, Day 1, Day 2, Day 7, Day 14
  Pharmacodynamic assessments in blood will be listed and summarized by dose level
Wound healing | Day 0, Day 1, Day 2, Day 7, Day 14, Day 60
  Assessment of wound healing scored according to a modified ASEPSIS method

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Memorial Health, Savannah, Georgia
  - Indiana University, Indianapolis, Indiana
  - Mayo, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - NYU Langone Health, New York, New York
  - Duke Cancer Center, Durham, North Carolina
  - MD Anderson Cancer Center, Houston, Texas
  - Audie Murphy VA, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No